CLINICAL TRIAL: NCT06896760
Title: A Mass Balance Study of [14C]ABSK011 in Healthy Adult Male Chinese Participants
Brief Title: A Mass Balance Study of [14C]ABSK011
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABSK-011-103
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]ABSK011 (Experimental): Participants will receive a single oral administration of approximately 200 mg/120 µCi [14C]ABSK-011 suspension after a low-fat breakfast on day 1 morning.
  Interventions: Drug: [14C]ABSK011

INTERVENTIONS:
Drug: [14C]ABSK011 — The standard meal was taken the night before administration, and the patient was fasted for at least 10 h without drinking water overnight. The next morning, eat a low-fat meal, finish the meal within 30 minutes, and take the test drug with warm water 30 minutes (±5 minutes) after the beginning of the meal. The total volume of warm water and suspension liquid is about 240 mL. Except for meals and administration, no water was allowed 1 hour before and 1 hour after medication. No food is allowed for 4 hours after taking the medication. Throughout the study, participants received meals provided by the center at approximately the same time each day.

SUMMARY:
This study is a single-site, open-label, single-cohort, single-dose study to assess the absorption, metabolism, and excretion profile of [14C] ABSK011 in healthy adult male subjects. The study plans to enroll 6 to 8 healthy male subjects to ensure at least 6 evaluable subjects.

DETAILED DESCRIPTION:
Participants will be screened no more than 14 days before the dose (D-14 through D-3) and admitted to the clinical trial unit 2 days before the dose (D-2). Participants will receive a single oral administration of approximately 200 mg/120 µCi [14C]ABSK-011 suspension after a low-fat breakfast on day 1 morning.

Urine and stool samples will be collected from participants before and at specified intervals between 0 and 192 hours after taking the drug and blood samples will be collected at specified time points between 0 and 120 hours before and after taking the drug.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who fully understand the content, procedures and possible adverse reactions before the study, and voluntarily sign the informed consent form, and can complete the study in accordance with the requirements in the protocol;
2. Healthy male participants aged 18 to 45 years (including 18 and 45 years) at screening;
3. Weight ≥ 50 kg, body mass index (BMI) between 19 and 26 (including 19 and 26), BMI = weight (kg)/height (m) ^2;
4. Participants must have regular defecation in the past three months;
5. Male participants of childbearing potential must agree to use effective contraceptive methods during the study and within 6 months after administration of study drug . Male subjects must agree to not donate sperm during this period.

Exclusion Criteria:

1. Abnormal and clinically significant complete physical examination, vital signs, digital rectal examination, laboratory tests (hematology, blood biochemistry, urinalysis, coagulation function, stool routine + occult blood, thyroid function, etc.), 12-lead electrocardiogram, chest X-ray (anteroposterior position), abdominal B ultrasound (hepatobiliary, pancreas, spleen and kidney);
2. Tested positive for any one of the following: serum hepatitis B surface antigen (HBsAg), hepatitis B e antigen (HBeAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antigen/antibody, treponema pallidum antibody (Syphilis) screening;
3. The baseline of heart rate corrected QT, QTcF interval prolongs ≥450ms; family history of long QT syndrome (Note: QTc interval is corrected by Fridericia formula);
4. Known or persistent mental disorders that may interfere with the subject's participation in the study, as judged by the investigator;
5. Known history of allergy to any drug or food;
6. Participants who have participated in drug trials within 3 months before dosing.
7. Participants who have participated in this study or any other study related to ABSK011, and have previously exposed to ABSK011;
8. Known history of drug abuse or tested positive in drug abuse screening;
9. Participants with any other factors that may influence the participation in the study, which may affect the subject's compliance with the protocol, interfere with the interpretation of the study results, or expose the subject to risk, as judged by the investigator.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-04-07 (Estimated); Primary Completion 2025-11-07 (Estimated); Study Completion 2026-04-07 (Estimated)

PRIMARY OUTCOMES:
Cumulative excretion rate of radioactivity in excreta (urine, feces) and total radioactivity (urine and feces) | All excreted urine and feces samples at specified time points during 0-192 hours after dosing will be collected.
  To assess the routes and rates of elimination of ABSK011 and its metabolites after single oral administration of [14C]ABSK011 in healthy adult male subjects
Percentage of each metabolite in urine and feces relative to the administered dose (% administered dose), or percentage of metabolites in plasma relative to total exposure AUC (% AUC); | Conduct testing within 1 month after all subjects collect plasma, urine, and fecal samplesat all time points required by the protocol
  To determine the metabolism and elimination pathways of ABSK011 after single oral administration of [14C] ABSK011 in healthy adult male subjects, and identify major metabolites.All excreted urine and feces samples at specified time points during 0-192 hours after dosing will be collected.
%AUC | Conduct testing within 1 month after all subjects collect all samples at all time points required by the protocol
  To evaluate the pharmacokinetics of ABSK011 and its major metabolites in the urine of healthy adult male subjects after a single oral administration [14C] of ABSK011.

SECONDARY OUTCOMES:
Frequency, type and severity of adverse events/serious adverse events; changes in vital signs, 12-lead ECGs, laboratory tests, etc. | From signing the ICF until 9 days after the first dosing
  To assess the safety and tolerability of a single oral dose of approximately [14C] ABSK011 in healthy adult male subjects

CONTACTS AND LOCATIONS:
Overall Officials: Quankun Zhuang, Doctor, Principal Investigator — Beijing GoBroad Hospital; Xuemei Liu, Doctor, Principal Investigator — Beijing GoBroad Hospital
Locations (1):
- Beijing GoBroad Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No